CLINICAL TRIAL: NCT02449005
Title: A Phase I/II Double-Blind Randomised Controlled Clinical Trial To Study The Safety and Efficacy Of A Novel Regenerative Treatment Of Infrabony Periodontal Defects Using Autologous Alveolar Bone-Marrow Mesenchymal Stem Cells (aBM-MSCs).
Brief Title: Autologous Alveolar Bone Marrow Mesenchymal Stem Cells for the Reconstruction of Infrabony Periodontal Defects
Acronym: PerioRegen
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Collaborators: University of Glasgow (Other)
Responsible Party: Principal Investigator, Danae A. Apatzidou, Assistant Professor, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ELKE-90467
Record Dates: First submitted 2015-05-13; First posted 2015-05-20 (Estimated); Last update posted 2022-06-03 (Actual); Status verified 2022-06

CONDITIONS: Chronic Periodontitis
Keywords: regeneration; stem cells; infrabony periodontal defect; fibrin glue; collagen fleece
MeSH Terms: conditions — Chronic Periodontitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The participant, care provider, investigator/outcome assessor is not aware of the treatment modality
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group A (Experimental): Group A (BM-MSCs/fibrin glue/collagen fleece) will receive regenerative treatment using autologous bone marrow mesenchymal stem cells free of animal derived reagents, produced in clean room facilities and seeded into collagen scaffolds enriched with autologous fibrin glue
  Interventions: Biological: BM-MSCs/fibrin glue/collagen fleece
- Group B (Experimental): in Group B (Fibrin glue/collagen fleece), a collagen fleece enriched with autologous fibrin glue devoid of stem cells will fill the osseous defect
  Interventions: Other: Fibrin glue/collagen fleece
- Group C (Active Comparator): Group C will receive open flap debridement retaining the soft tissue wall of the pocket
  Interventions: Procedure: Open flap debridement

INTERVENTIONS:
Biological: BM-MSCs/fibrin glue/collagen fleece — Xeno-free, clinical-grade, autologous alveolar bone marrow mesenchymal stem cells enriched with autologous fibrin glue and loaded into a commercially available collagen fleece.
  Arms: Group A
Other: Fibrin glue/collagen fleece — The biocomplex of autologous fibrin glue and collagen fleece devoid of stem cells will fill the osseous defect
  Other Names: Procedure/Surgery/Growth factors
  Arms: Group B
Procedure: Open flap debridement — Group C will receive minimally invasive surgery employing papilla preservation techniques in addition to retaining the soft tissue wall of the pocket. There will be no use of grafting materials
  Arms: Group C

SUMMARY:
Systemically healthy periodontitis patients are recruited from new referrals to the Department of Periodontology and Biology of Implants, AUTh. After completion of non-surgical periodontal treatment those subjects who have at least one interdental osseous defect with probing pocket depth and clinical attachment level of ≥ 6mm and an intrabony component of ≥ 3mm with no endodontic or furcation involvement are randomly allocated into one of the three treatment groups. Group A receives regenerative treatment using autologous bone marrow mesenchymal stem cells free of animal derived reagents, produced in clean room facilities and seeded into collagen scaffolds enriched with fibrin glue; in Group B, a collagen fleece enriched with fibrin glue devoid of stem cells fills the osseous defect; Group C receives open flap debridement retaining the soft wall of the defect. Thereafter, subjects are followed for 12 months and are repeatedly assessed based on clinical, radiographic, immunological and microbiological parameters.

In a series of cases, tissue engineering in a similar manner to Group A will be applied to treat isolated periodontal interdental defects, in combination with the novel "closed surgical technique".

DETAILED DESCRIPTION:
Aims & Objectives The present study describes a novel method to regenerate periodontal tissues in periodontal infrabony defects using autologous BM-MSCs, free of animal derived reagents, produced in clean room facilities enriched with autologous fibrin glue and seeded into commercially available collagen scaffolds (collagen fleece).

Primary objective This study aims to assess the efficacy of a novel regenerative treatment of periodontal infrabony defects using a biocomplex of BM-MSCs/fibrin glue/collagen fleece, as compared to a cell-free grafting substitute of fibrin glue/collagen fleece and to a control treatment approach of open flap debridement with no adjunctive use of grafting materials.

Secondary Objectives

* To document the stability of the enhanced treatment outcome and to continue to assess the safety and effectiveness of BM-MSCs transplantation as compared to the control treatment of open flap debridement over the study period.
* Determine the immunological and microbiological profiles of the participants throughout the study period in an attempt to understand local and systemic effects of the transplantation of BM-MSCs in chronically diseased sites, such as the infrabony periodontal defect. In addition, the healing response to treatment will be determined throughout the observation period (baseline to 12-months).

Study Design

Investigational products aBM-MSCs cultures will be established from osseous biopsies derived from bone marrow of the alveolar bone in each patient belonging to Group A. Briefly, after a thorough oral rinse with chlorhexidine 0.12% for 1min, an osteotomy using a trephine drill will be performed in the alveolar bone and a 2x8 mm osseous core will be harvested. The area will be irrigated with saline solution and then flaps will be sutured to achieve primary closure at the donor site. The bone sample will be then immediately placed in sterile tubes containing HBSS and antibiotics/antimycotics and will be transported to a Good Laboratory Practice (GLP)-compliant authorized facility meeting the quality guidelines set by the European Union for the preparation of clinical-grade stem cell cultures for delivery to the patient. aBM-MSC isolation will be performed using the enzymatic dissociation method, as previously described (Bakopoulou 2013). For culture expansion, autologous serum obtained from 60ml of venous blood collected from each subject will be used to supplement aMEM cell culture medium, in order to avoid the use of any animal derived reagents, such as bovine serum. The osseous biopsy will be immediately processed to ensure high viability of the established cultures. After expansion for two passages (approximate time needed 16-24 days depending on cell donor) cells will be harvested for delivery to the patient. For cell dissociation and passaging, highly purified, GMP compatible recombinant enzymes (Tryple, Thermo Fisher Scientific) will be used to avoid use of porcine trypsin. At this stage, a sample of 20ml venous blood will be required for the preparation of the autologous fibrin glue in Group B, as in Group A initial bloodletting (60ml) will cover the needs of the cell cultures and fibrin glue preparation. Subsequently, fibrin glue will be loaded with- (Group A) or without- (Group B) stem cells into a commercially available collagen fleece scaffold directly before clinical application.

Quality control of the established BM-MSC cultures before clinical application

Before delivery to the patient, all BM-MSCs cultures will be evaluated for:

* Viability using Trypan Blue exclusion
* Sterility: cultures will be tested for potential contamination from bacteria, mycoplasma and endotoxins (LAL test)
* "Stemness" properties based on the minimal criteria established by the International Society for Cellular Therapy (ISCT) regarding MSCs (Dominici et al 2006).

Note: Methodology on stem cell characterization methods is analytically described in previous publications by our research group (Bakopoulou et al. 2013).

After application of the BM-MSCs/fibrin glue/CaCl2 mixture into the collagen scaffolds, a small sample of the biocomplex of randomly selected cases will be separated using surgical scissors and will be transferred to the lab for further (in parallel to the clinical application) ex vivo characterization of stem cell behavior in a biomimetic microenvironment. This will allow correlation between stem cell behavior and the clinical outcome, since retrieval and analysis of the regenerated tissues directly from the host is not feasible for ethical reasons.

Preparation of autologous fibrin glue Twenty ml of venous blood will be collected from the ante-cubital fossa of patients in Groups A and B and blood samples will be immediately transferred to a falcon tube, which contains anticoagulant. After determination of the platelet counts the blood sample will be centrifuged (2000rpm, 10min) and plasma will be separated and stored in another falcon. Platelets counts will be then determined and the sample will be centrifuged again. PRP (platelet rich plasma containing 1,000,000 plts/ul) will be then separated from the supernatant PPP (platelet poor plasma) and both preparations will be further processed following a standard protocol for fibrin glue preparation (Biohellenika, Thessaloniki, Greece).

Design of the clinical arm of the study

Pre-selection of Subjects Subjects will be recruited from new referrals at the Department of Preventive Dentistry, Periodontology and Implant Biology; no external advertising or recruitment will be undertaken. Subjects will be in good general health.

Admission into the Study Before admission into the study, each subject will be informed by the principal investigator of the nature and risks of the study both orally and in writing (Subject Information Form) and written informed consent (Subject Informed Consent Signature Form) will be obtained. Each subject will be given a copy of their duly signed consent form to maintain for their own records. The subjects' personal demographics and medical history and study suitability in accordance with the inclusion and exclusion criteria set in the protocol will be recorded. Subjects may continue any medications not included in the exclusion criteria; however, these medications should be documented together with any concurrent medical condition not pre-excluded.

Procedures for Subject Withdrawal or Discontinuation Any subject, who wishes to withdraw from the study for personal or any other reason, is entitled to do so. However, the reason for the withdrawal of any subject from the study in addition to whether the reason is related to the test product will be recorded by the principal investigator. Any participant failing to attend more than twice is removed from the study. Subjects that experience an adverse event will be excluded from further participation in the study.

If a subject wishes to withdraw from the study, all efforts will be made to complete and report the observations as thoroughly as possible up to the date of withdrawal. Subjects will be asked to consider giving further information as to the reason(s) for the withdrawal. Any information reported will be recorded.

Expected Duration of each subject participation Each subject is expected to attend nine visits in total over a period of 12 months; one screening visit, one treatment visit to receive surgical treatment of the designated area, four follow-up reviews and three additional visits for clinical and radiographic reassessment and sample collection (whole saliva, gingival crevicular fluid (GCF), subgingival plaque).

Investigators' calibration and randomisation Patients will be screened for eligibility by one examiner and will be enrolled one at a time on a continuous basis after obtaining a code number. A trial contributor not involved in data collection will perform the randomisation and announce the treatment modality to the therapist using telephone communication. Clinical assessments will be carried out by a single examiner who will have no access to previous recordings and is not otherwise involved in other clinical procedures. An investigator calibration exercise will be performed to obtain acceptable intra-examiner reproducibility for PPD, CAL, and evaluation of defect anatomy. Intra-examiner reproducibility will be evaluated by Intraclass Correlation Coefficient (ICC) and Bland-Altman 95% limits of agreement (Bland and Altman, 1999).

Statistical analysis of experimental data The analysis will be performed using the IBM Statistics SPSS 20.0, software. Data will be expressed as means +/- standard deviation (SD). Unbalances between the test and control groups that are generated by the randomisation procedures will be assessed using the independent samples t-test for continuous variables and the Fisher's Exact test or the Chi-Square test for categorical variables. The significance of the treatment effects on the dependent variables CAL changes, PPD changes and radiographic changes will be estimated by constructing linear mixed models using the SPSS MIXED procedure. For all analyses the statistical significance will be set at p<0.05.

Ethical considerations / Authorisations for stem cell cultures Biohellenika, Thessaloniki, Greece provides state of the art facilities and labs that are operating under the strictest regulations for stem cells processing and storage. The labs are licensed according to Government's order 26/24-3-2008 (regulation of Greek law according to European law 2004/23/K of and Council 31-3-2004 for the establishment prototypes of quality and safety for the donation, the purchase, the quality controls the cryopreservation, storage and the distribution of human tissues and cells (EEL 102/7-4-2004) and the related guidelines 2006/17 EK (EEL 38/9/2006) and 2006/86EK (EEL 294/25-10-2006). The license F 6172/17514/1269 is published in Gov. paper 2589 31/12/2009.

Since November 2014, Biohellenika operates under the new law 3984, published in Gov paper No 150, 2011 after a positive recommendation of the National Transplant Committee to Department of Health and at the moment the new license is about to published in the Gov paper.

The labs and the procedures are accredited by the American Association of Blood Banks (AABB), last inspection 30th of September, 2014 and by the National System of Accreditation according to ISO 15189:2007. Also the labs are certified according to ISO 9001:2008, for processing, quality control and cryopreservation of autologous cell lineages and ISO 13485:2003 for the cryopreservation system which is also an international patent of Biohellenika.

Clean rooms operate according to the guidelines of BSR Ingenieur-Buro with ISO 14644-5. The security levels meet all the standards ISO 27001 and the company is licensed and regulated by the Data Protection Authority.

The labs are surveyed 24 hours for air quality and equipped with Cryo-View data base System, ISBT 128 barcoding system, Temperature -Liquid N2 level, Security Alarms and two power generators.

Study Schedule Clinical design and interventions for autologous transplantation of BM-MSCs Subjects with severe chronic periodontitis will be scheduled to receive non-surgical periodontal treatment under local anaesthesia using hand and power driven instruments, in addition to motivation in periodontal care and thorough oral hygiene instructions. Subjects will be clinically reassessed six weeks after the completion of non-surgical treatment and those subjects with remaining periodontal pockets (PPD & CAL ≥ 6mm; infrabony component ≥ 3mm) and no overt signs of gingival inflammation will be screened for suitability to participate in the current study. The screening visit will include an initial full-mouth periodontal examination, intra-oral radiographic examination and fulfilment of inclusion/exclusion criteria. In case of suitability, the nature of the study will be explained in detail to all subjects and a signed consent form approved by the Ethics Committee of the Dental School, AUTh. will be obtained from each participant. Then, patients will be randomly allocated into one of the three treatment Groups (-A, -B and -C). A single defect will be treated in each patient.

Subsequently, an osseous biopsy and blood samples will be collected from the participants of Group A under strict sterile conditions. Each sample will be then immediately placed in sterile tubes and will be transported to Biohellenika, Thessaloniki, Greece (http://www.biohellenika.gr) for stem cell isolation and expansion according to a strict protocol (Bakopoulou et al. 2013, Bakopoulou et al. in preparation). Since MSCs will be isolated and expanded in vitro in GLP-class clean rooms meeting the quality guidelines set by the European Union and no animal derived reagents will be used throughout the experiments for autologous transplantation, the cells are considered safe for human clinical cell therapy applications. In Biohellenika facilities 60ml of venous blood will be collected from each subject in Group A shortly after the biopsy harvest, so that autologous serum is used for the isolation and culture expansion of the autologous stem cells. In addition, autologous fibrin glue will be used to load the BM-MSCs onto the collagen fleece. In addition, a blood sample of 20ml will be collected from subjects in Group B, in order to provide fibrin glue which will enrich the collagen fleece before surgical placement into the osseous defect. Finally, subjects in Group C will not be called for bloodletting as the infrabony defects in these individuals will be surgically managed by open flap debridement with no adjunctive use of grafting materials.

As part of the GLP quality control, the MSCs will be analysed for sterility and endotoxins and will be also tested for potential contamination from bacteria (BD BACTEC™), mycoplasma and endotoxins (LAL test).

Local anaesthesia (1.8ml of 2% lidocaine with 1:80,000 epinephrine; Lignospan special, Septodont) will be infiltrated in the buccal and lingual aspects of the involved teeth avoiding the papillae. Then, strictly intra-sulcular incisions will be performed to preserve the gingival tissues and in particular the interdental papilla associated with the bone-dental defect (Cortellini, 2012; Cortellini and Tonetti 2007). The defect will be debrided and the root will be carefully planed with the combined use of Gracey curettes and power-driven instruments (EMS Piezon®, EMS, Nyon, Switzerland). Care will be taken to retain the soft-tissue wall of the defects and the osseous defect will be irrigated with saline to control bleeding.

In Group A, the grafting material (BM-MSCs enriched with fibrin glue) will be delivered in two insulin syringes each containing 5x10E6 cells/100μl fibrin and will be gently loaded onto the collagen fleece and polymerized with the addition of CaCl2. Subsequently, the biocomplex will be gently packed into the defect until complete fill. Handling of the scaffold is done with care to avoid any destruction of viable cells.

In Group B, the collagen fleece enriched with fibrin glue devoid of viable cells will fill the vertical bone defect with caution. In Groups -A and -B the delivery of fibrin glue with/without viable cells will be identical, so that the therapist is blinded to the procedures.

Group C, patients will receive open flap debridement and root planing of the root surface in a similar manner as subjects in Groups -A and -B, but there will be no adjunctive use of grafting materials.

The operator will be blinded to the treatment modality (Groups -A and -B), while in Group C since no grafting materials will be used, the treatment modality will become obvious to the operator but this will take place towards the conclusion of the surgery, after the collection of clinical data. Papilla preservation techniques and minimally invasive surgical techniques will be sought in all groups, avoiding scoring the periosteum. Flaps will be repositioned and sutured using a single modified internal mattress suture (5-0 Monosyn, Braun) at the defect-associated interdental area and similar sutures will be employed to close the flaps in any other interdental areas. Two weeks post-surgery clinical observation for uneventful healing or presence of adverse tissue reaction will be performed followed by suture removal.

Case series for tissue engineering In a series of cases (five) having similar inclusion/criteria as above but without going through randomisation tissue engineering is applied following the same methodology as in Group A. In theses cases, the tissue engineered construct (biocomplex) is applied to treat isolated interdental periodontal defects using a newly designed surgical technique the so-called "closed surgical technique". In brief, this technique entails retraction of gingival flaps in a closed manner without dissecting the soft-tissues or the interdental papilla. This technique minimises tissue trauma, postoperative discomfort and enhances soft-tissue aesthetics.

Post-operative care Post-operative pain will be controlled with Ibuprofen (600mg) at the end of the surgical procedure and 12h later if in pain. Amoxicillin (500mg / 8 hours for five days) will be prescribed to all participants. All patients will be instructed to use 0.12% chlorhexidine twice daily and avoid brushing, flossing and chewing hard in the treated area for four weeks. During this 4-week period, stringent post-operative supportive program care will be instituted at bi-weekly intervals, and after that patients will discontinue rinsing with chlorhexidine solution and resume oral hygiene. Interdental cleaning will commence six weeks post-surgery for all Groups. Thereafter, subjects will be seen at three, six and 12 months for periodontal supportive care.

Clinical recordings Full-mouth and site-specific periodontal recordings including BOP; Plaque Index (presence/absence of plaque); PPD and CAL will be determined using a manual periodontal probe (Hu-Friedy XP-23/QW) to the nearest millimetre at six sites per tooth and parallel to the long axis at four time-points; baseline, 6-, 9-, 12-months. Clinical measurements at the designated sites (infrabony defects) will be determined prior to surgery and before anaesthesia (baseline). Intra-surgical assessments will be carried out once during surgery.

Intra-surgical clinical assessments The defect morphology (one-, two-, three-walls or combination) will be determined intra-surgically by the number of bone walls associated with the lesion; The distance between the cemento-enamel junction and the bottom of the defect (CEJ-BD) will be determined in mm; The distance from the CEJ to the most coronal interproximal level of the bone crest (CEJ-BC) will be determined in mm; The total defect depth: the distance between the bone crest and the bottom of the defect (BC-BD) will be determined in mm; The width of the defect width (horizontal distance between the bone crest and the root surface) will be determined in mm.

If the CEJ is not detectable due to a cervical restoration the restoration margin (RM) will serve as reference point for clinical and radiographic measurements.

Radiographic evaluation Intraoral digital radiography will be utilised to determine the bone regeneration of the infrabony defects at six time points; baseline, 6-weeks, 3-, 6-, 9-, 12-months. Standardised periapical digital radiographs (RadioVisioGraphy; Trophy Radiology S.A., Paris, France) will be obtained using the long-cone paralleling technique. To standardise the exposure geometry, a customised bite-block of an elastic impression material will be adjusted on the sensor holder, stored in sealed plastic containers at room temperature and will be reused during every recall radiographic appointment.

In a similar manner as the intra-surgical assessment, the following anatomical landmarks will be defined on the x-rays: the cementoenamel junction (CEJ), the most coronal level of the alveolar bone (BC) and the apical extent of bone loss (BD). In more detail, the location of the CEJ will be identified; the most coronal area where the periodontal ligament retains an even width will be identified on the radiograph to indicate the most apical extension of bone loss. The infrabony defect will be calculated by measuring the width of the defect at the most coronal aspect and at the base; the distance between CEJ-BD and BC-BD; the distance between CEJ-BC; the angle between the vertical axis of the root and the interdental bone wall (Tonetti et al. 1993). Radiographic evaluation of bone regeneration will be defined on a high definition monitor by the same calibrated examiner who is blinded to the treatment modality and does not have access to previous recordings. Assessments will be carried out using the measurement tool for numerical measurements (VixWin™ Platinum|Gendex software) with reference to a metal bar of standard length (5mm) that will be attached onto the sensor.

Collection of specimens Samples will be collected in the following order at six time points; baseline, 6-weeks, 3-, 6-, 9-, 12-months.

(i) Saliva Saliva will be collected prior to clinical periodontal measurements or any periodontal intervention and generally in the morning following an overnight fast during which subjects are requested not to drink (except water) or chew gum. Whole saliva samples will be obtained by expectorating into 30ml polypropylene tubes for 5 minutes.

(ii) GCF Gingival crevicular fluid samples will be obtained from the buccal interdental aspects of the defects. Before GCF collection, the surfaces will be gently air dried and isolated from saliva by placing cotton rolls and using a saliva ejector. Then, supragingival plaque will be carefully removed with sterile curettes and paper strips (Periopaper, OraFlow Inc., Smithtown, NY, USA) will be placed in the periodontal pocket until mild resistance is felt for 30s. Care will be taken to avoid mechanical trauma when placing the strips and those strips contaminated with blood will be discarded. Each strip per patient will be stored in a separate 1.5ml micro-centrifuge tube, and stored at -70°C. Prior to use, the proteins on the strips will be eluted into 500µl of phosphate buffered saline (PBS) supplemented with BSA (1% v/v).

(iii) Plaque Following GCF collection, subgingival plaque will be collected from the designated site. The sampling area will be isolated from saliva, gently dried with air, and after ensuring that no supragingival plaque deposits are present two paper points will be placed for 30s into the periodontal pocket and a pooled sample will be collected. All samples will be stored in Eppendorf tubes (Eppendorf, Hamburg, Germany) at -80°C before processing. Paper points will be used for the collection of microbial plaque in order to avoid mechanical disturbance of the periodontal tissues.

Data management The investigators must ensure that the subject's anonymity is maintained. On any study-related documentation, subjects should only be identifiable by their initials, gender, and/or subject number. Personal information (i.e. medical cards) will be kept in a separate, secure location, away from other study specific data with restricted access to the principal investigator only.

Informed consent process It is the responsibility of the principal investigator to obtain in writing consent from the subject. The informed consent form will consist of two separate documents; a Subject Information Form and a Subject Informed Consent Signature Form; both documents will be approved by the Ethical committee of the Dental School, AUTh prior to the study. The subject information form will provide an adequate explanation, in native non-technical language that is understandable to the subject, of the aims, objectives, methods, anticipated benefits and potential hazards of the study. The principal investigator must then provide ample time for the subject to read and understand the informed consent form and to consider participation in the clinical investigation. The principal investigator and the subject must both sign and date the form before the subject can participate in the clinical investigation. Each subject will then be issued with a copy of their duly signed and dated informed consent form and any other written information.

ELIGIBILITY:
Inclusion Criteria:

* Following non-surgical periodontal treatment, advanced chronic periodontitis patients, who are able to maintain plaque scores of less than 25% and have at least one deep infrabony defect with PPD and CAL of ≥ 6mm and an infrabony component of ≥ 3mm with no endodontic or furcation involvement as detected on the radiographs will be scheduled for surgery and will be followed for 12 months.

Exclusion Criteria:

* Exclusion criteria: poorly controlled systemic disease, heavy smoking (>20cigs/day), drug induced gingival hyperplasia, bisphosphonate medication, anti-inflammatory drugs, bone metabolic diseases or disorders that compromise wound healing, immunosuppressive therapy or radiation, alcohol intake, drug abuse over the past year, significant concurrent illness, pregnancy/lactation, poor compliance during the initial phase of treatment, compromised oral hygiene (PI ≥25%).

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
A reduction in the distance in mm from the bottom of the periodontal pocket to the cementoenamel junction using a manual probe (Hu-Friedy XP-23/QW, Hu-Friedy, Chicago, IL, USA) with 20-25g of pressure by a single calibrated examiner. | up to 12- months
  Clinical data (gain in clinical attachment level (CAL))

SECONDARY OUTCOMES:
A reduction in the distance in mm between the gingival margin and the bottom of the defect using a manual periodontal probe (Hu-Friedy XP-23/QW) by a single calibrated examiner. | up to 12-months (baseline, 6-, 9-, 12- months)
  Clinical data (reduction in probing pocket depth (PPD))

OTHER OUTCOMES:
A change in the distance in mm between the cementoenamel junction and the bottom of defect will be determined using a single evaluator. | Baseline, 6-weeks & 3-, 6-, 9-, 12- months
  Radiographic data (CEJ-BD change)
A change in the distance in mm between the bone crest to bottom of defect will be determined using a single evaluator. | Baseline, 6-weeks & 3-, 6-, 9-, 12- months
  Radiographic data (BC-BD change)
Composite measure of biomarkers will be examined to evidence the healing and immune response during the observation period | Baseline, 6-weeks & 3-, 6-, 9-, 12- months
  Immunological data; changes
Clinical measurements after surgical debridement of the area will determine the morphology of the osseous defect | Baseline
  Intrasurgical clinical data (CEJ-BD; BC-BD; width of the defect; number of bone walls)

CONTACTS AND LOCATIONS:
Overall Officials: Antonis Konstantinidis, Professor, Study Chair — Dept. of Periodontology and Implant Biology, School of Dentistry, Aristotle University of Thessaloniki
Locations (1):
- Dental School, Aristotle University, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bakopoulou A, Leyhausen G, Volk J, Koidis P, Geurtsen W. Comparative characterization of STRO-1(neg)/CD146(pos) and STRO-1(pos)/CD146(pos) apical papilla stem cells enriched with flow cytometry. Arch Oral Biol. 2013 Oct;58(10):1556-68. doi: 10.1016/j.archoralbio.2013.06.018. Epub 2013 Jul 18. PMID 23871383
- [Background] Bland JM, Altman DG. Measuring agreement in method comparison studies. Stat Methods Med Res. 1999 Jun;8(2):135-60. doi: 10.1177/096228029900800204. PMID 10501650
- [Background] Cortellini P, Tonetti MS. Minimally invasive surgical technique and enamel matrix derivative in intra-bony defects. I: Clinical outcomes and morbidity. J Clin Periodontol. 2007 Dec;34(12):1082-8. doi: 10.1111/j.1600-051X.2007.01144.x. Epub 2007 Oct 22. PMID 17953696
- [Background] Cortellini P. Minimally invasive surgical techniques in periodontal regeneration. J Evid Based Dent Pract. 2012 Sep;12(3 Suppl):89-100. doi: 10.1016/S1532-3382(12)70021-0. PMID 23040341
- [Background] Dominici M, Le Blanc K, Mueller I, Slaper-Cortenbach I, Marini F, Krause D, Deans R, Keating A, Prockop Dj, Horwitz E. Minimal criteria for defining multipotent mesenchymal stromal cells. The International Society for Cellular Therapy position statement. Cytotherapy. 2006;8(4):315-7. doi: 10.1080/14653240600855905. PMID 16923606
- [Background] Altman DG. Statistics in the medical literature: 3. Stat Med. 1999 Feb 28;18(4):487-90. doi: 10.1002/(sici)1097-0258(19990228)18:43.0.co;2-j. No abstract available. PMID 10070688
- [Derived] Apatzidou DA, Iliopoulos JM, Konstantinidis A, Verma M, Hardy P, Lappin DF, Nile CJ. Inflammatory and bone remodelling related biomarkers following periodontal transplantation of the tissue engineered biocomplex. Clin Oral Investig. 2024 Jun 7;28(7):361. doi: 10.1007/s00784-024-05754-8. PMID 38847929
- [Derived] Apatzidou DA, Bakopoulou AA, Kouzi-Koliakou K, Karagiannis V, Konstantinidis A. A tissue-engineered biocomplex for periodontal reconstruction. A proof-of-principle randomized clinical study. J Clin Periodontol. 2021 Aug;48(8):1111-1125. doi: 10.1111/jcpe.13474. Epub 2021 May 14. PMID 33899259